CLINICAL TRIAL: NCT02044822
Title: A Phase 2, Single Arm Study Evaluating the Efficacy and Safety of Idelalisib in Combination With Rituximab in Patients With Previously Untreated Chronic Lymphocytic Leukemia With 17p Deletion
Brief Title: Efficacy and Safety of Idelalisib in Combination With Rituximab in Patients With Previously Untreated Chronic Lymphocytic Leukemia With 17p Deletion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-312-0133; 2013-003314-41 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2017-03

CONDITIONS: B-cell Chronic Lymphocytic Leukemia (CLL) With 17p Deletion
Keywords: Chronic Lymphocytic Leukemia; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — idelalisib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Idelalisib + rituximab (Experimental): Participants will receive rituximab for 8 weeks and Idelalisib continuously throughout the study (up to 10 years).
  Interventions: Drug: Idelalisib; Drug: Rituximab

INTERVENTIONS:
Drug: Idelalisib — 150 mg tablets administered orally twice daily
  Other Names: GS-1101; CAL-101; Zydelig®
Drug: Rituximab — 375 mg/m^2 administered intravenously once weekly x 8 weeks
  Other Names: Rituxan

SUMMARY:
The primary objective of this study is to evaluate overall response rate (ORR) following treatment with idelalisib plus rituximab in participants with previously untreated chronic lymphocytic leukemia (CLL) with 17p deletion.

An increased rate of deaths and serious adverse events (SAEs) among participants with front-line CLL and early-line indolent non-Hodgkin lymphoma (iNHL) treated with idelalisib in combination with standard therapies was observed by the independent data monitoring committee (DMC) during regular review of 3 Gilead Phase 3 studies. Gilead reviewed the unblinded data and terminated those studies in agreement with the DMC recommendation and in consultation with the US Food and Drug Administration (FDA). All front-line studies of idelalisib, including this study, were also terminated.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented diagnosis of B-cell CLL, according to International Workshop on Chronic Lymphocytic Leukemia 2008
* Presence of 17p deletion in CLL cells as demonstrated by fluorescence in-situ hybridization (FISH) testing
* No prior therapy for CLL other than corticosteroids for disease complications
* CLL that warrants treatment
* Presence of measurable lymphadenopathy
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Key Exclusion Criteria:

* Known histological transformation from CLL to an aggressive lymphoma (ie, Richter transformation)
* Known presence of myelodysplastic syndrome
* History of a non-CLL malignancy except for the following:

  * the malignancy has been in remission without treatment for ≥ 5 years prior to enrollment, or
  * carcinoma in situ of the cervix, or
  * adequately treated basal or squamous cell skin cancer or other localized non-melanoma skin cancer, or
  * asymptomatic prostate cancer without known metastatic disease and with no current requirement for therapy or requiring only hormonal therapy and with normal prostate specific antigen for ≥ 1 year prior to enrollment, or
  * ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone, or
  * other adequately treated Stage 1 or 2 cancer currently in complete remission
* Evidence of ongoing systemic bacterial, fungal, or viral infection at the time of enrollment
* Ongoing liver injury
* History of noninfectious pneumonitis
* Ongoing inflammatory bowel disease
* History of prior allogeneic bone marrow progenitor cell or solid organ transplantation
* Ongoing immunosuppressive therapy other than corticosteroids
* Received last dose of study drug on another therapeutic clinical trial within 30 days prior to enrollment
* Prior or ongoing clinically significant illness, medical condition, surgical history, physical finding, electrocardiogram (ECG) finding, or laboratory abnormality

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2016-04-27 (Actual); Study Completion 2016-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (56):
- United States (11):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Innovative Clinical Research Institute, Whittier, California
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - The University of Chicago Medicine, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University, Durham, North Carolina
  - GHS Cancer Institute, Greenville, North Carolina
  - Compass Oncology, Portland, Oregon
  - Willamette Valley Cancer Center and Research Institute, Springfield, Oregon
  - Hospital of the University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
- Australia (5):
  - St Vincent's Hospital, Sydney, Darlinghurst, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - St Vincent's Hospital, Melbourne, Fitzroy, Victoria
  - Liverpool Hospital, Liverpool
- Austria (3):
  - Innsbruck University Hospital, Inner Medicine,, Innsbruck
  - Univ. Klinik für Innere Medizin III LKH, Salzburg
  - Medizinische Universität Wien, Univ. Klinik f. Innere Med. I, Abteilung für Hämatologie und Hämostaseologie, Vienna
- Belgium (2):
  - AZ Sint-Jan AV Brugge-Oostende, Bruges
  - University Hospital Leuven, Leuven
- Czechia (6):
  - University Hospital, Brno
  - Faculty Hospital Hradec Kralove, Hradec Králové
  - Hemato-Onkologicka Klinika Fn, Olomuc
  - Faculty hospital Ostrava, Ostrava-Poruba
  - Faculty Hospital Kralovske Vinohrady, Prague
  - Vseobecna Fakultim Nemocnice, Prague
- Aalborg University Hospital, Aalborg, Denmark
- France (4):
  - Centre Hospitalier Universitaire Hôpital Avicenne, Bobigny
  - CHRU de Lille, Hopital Claude Huriez, Lille
  - Centre Hospitalier Universitaire Nancy, Nancy
  - Hopital Pitie-Salpetriere, Paris
- University of Debrecen HSC Institute of internal Medicine, Department of Hematology, Debrecen, Hungary
- Italy (5):
  - Institute of Hematology "L. e A. Seràgnoli", Bologna
  - A.O.Spedali Civili Brescia, Brescia
  - A.O.Niguarda Ca' Granda, Milan
  - Azienda Ospedaliero Universitaria Policlinico di Modena, Modena
  - SCDU Medicina II ed Ematologia, A.O.U. San Luigi Gonzaga, Orbassano
- Poland (6):
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Szpital Specjalistyczny w Brzozowie, Brzozów
  - Malopolskie Centrum Medyczne s.c., Krakow
  - Wojewodzki Szpital Specjalistyczny, Lodz
  - Centrum Onkologii-Instytut Marii Sklodowskiej -Curie klinika Nowotworow Ukladu Chlonnego, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny, Wroclaw
- Portugal (2):
  - Centro Hospitalar De Lisboa Norte, E.P.E. - Hospital Santa Maria, Lisbon
  - IPO Porto Francisco Gentil, E.P.E, Porto
- Romania (3):
  - Emergency County Clinical Hospital Brasov, Brasov
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Regional de Oncologie Iasi, Iași
- Spain (4):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Clinic, Barcelona, Catalonia
  - Hospital Universitario Puerta De Hierro, Madrid
  - Hospital Clinico Universitario De Valencia (Chuv), Valencia
- United Kingdom (3):
  - Saint James's University Hospital, Leeds
  - Royal Liverpool & Broadgreen Univ. Hospitals, Liverpool
  - University Hospital Southampton NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe, and the United States. The first participant was screened on 06 August 2014. The last study visit occurred on 17 May 2016.
Pre-assignment Details: 130 participants were screened.
Groups:
- Idelalisib + Rituximab: Idelalisib (Zydelig®) 150 mg tablet twice daily + rituximab 375 mg/m^2 intravenously once weekly for 8 weeks
Period: Overall Study
Arm/Group | Idelalisib + Rituximab
Started | 102
Completed | 9 (Completed = reached primary efficacy endpoint of progressive disease or death.)
Not Completed | 93
Not completed — Study Terminated by Sponsor | 77
Not completed — Investigator's Discretion | 10
Not completed — Withdrew Consent | 3
Not completed — Initiation of Anti-Neoplastic Therapy | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set: participants who received at least 1 dose of study treatment
Groups:
- Idelalisib + Rituximab: Idelalisib 150 mg tablet twice daily + rituximab 375 mg/m^2 intravenously once weekly for 8 weeks
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black or African American | 2
  White | 94
  Not Permitted | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 91
  Not Permitted | 5
Region of Enrollment [Number; unit: participants]
  Romania | 4
  Hungary | 2
  United States | 19
  United Kingdom | 11
  Portugal | 2
  Spain | 7
  Austria | 3
  Czech Republic | 9
  Belgium | 2
  Denmark | 1
  Poland | 15
  Italy | 14
  Australia | 6
  France | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) was defined as the proportion of participants who achieve a confirmed complete or partial response. ORR was to be assessed by an independent review committee (IRC).
Population: Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Duration of Response
Description: Duration of response (DOR) was defined as the interval from the first documentation of confirmed complete response or partial response (by IRC) to the first documentation of definitive disease progression or death from any cause. Definitive disease progression is chronic lymphocytic leukemia (CLL) progression based on standard criteria, excluding lymphocytosis alone.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

3. Secondary Outcome: Nodal Response Rate
Description: Nodal response rate was defined as the proportion of participants who achieve a 50% decrease from baseline in the sum of the products of the greatest perpendicular diameters of index lesions. Nodal response rate was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

4. Secondary Outcome: Complete Response Rate
Description: Complete response rate was defined as the proportion of participants who achieve a confirmed complete response. Complete response rate was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the interval from first dose of study drug to the first documentation of definitive disease progression or death from any cause. Definitive disease progression is CLL progression based on standard criteria, excluding lymphocytosis alone. PFS was to be assessed by an IRC.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the interval from the start of study treatment to death from any cause.
Population: Due to the early termination of the study, efficacy data were not mature for all participants, and therefore the prespecified analyses were not conducted.
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

7. Secondary Outcome: Minimal Residual Disease Negativity Rate at Week 36
Description: Minimal residual disease (MRD) negativity rate was defined as the proportion of participants with MRD < 10^-4 assessed by flow cytometry in bone marrow at Week 36 after therapy initiation. For participants receiving the final dose of rituximab after the original scheduled date, the MRD assessment will be performed no fewer than 12 weeks after the last dose of rituximab.
Population: as for outcome 1
Arm/Group | Idelalisib + Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 17 months plus 30 days
Description: Intent-to-Treat Analysis Set
Arm/Group | Idelalisib + Rituximab
Serious Adverse Events (participants affected / at risk) | 46/102
Other Adverse Events (participants affected / at risk) | 98/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=102)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 6
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Glossitis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oral mucosal eruption (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Malaise (General disorders) | 1
Pyrexia (General disorders) | 11
Appendicitis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Cytomegalovirus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Intestinal sepsis (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Lower respiratory tract infection fungal (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Pneumocystis jirovecii infection (Infections and infestations) | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia influenzal (Infections and infestations) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Pneumonia pseudomonal (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Body temperature increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Transaminases increased (Investigations) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysgeusia (Nervous system disorders) | 1
Facial nerve disorder (Nervous system disorders) | 1
Confusional state (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Idelalisib + Rituximab (N=102)
Anaemia (Blood and lymphatic system disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 36
Dyspepsia (Gastrointestinal disorders) | 8
Mouth ulceration (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 17
Asthenia (General disorders) | 15
Chills (General disorders) | 13
Fatigue (General disorders) | 16
Oedema peripheral (General disorders) | 11
Pyrexia (General disorders) | 24
Bronchitis (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 10
Oral candidiasis (Infections and infestations) | 6
Respiratory tract infection (Infections and infestations) | 6
Upper respiratory tract infection (Infections and infestations) | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 6
Alanine aminotransferase increased (Investigations) | 39
Aspartate aminotransferase increased (Investigations) | 22
Transaminases increased (Investigations) | 6
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 8
Headache (Nervous system disorders) | 10
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 28
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 7

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, efficacy data were not available for all participants, and therefore the prespecified analyses were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years